CLINICAL TRIAL: NCT01613768
Title: Phase II Trial of Eribulin for Locally Advanced Refractory or Metastatic Salivary Gland Cancers
Brief Title: Eribulin Mesylate in Treating Patients With Recurrent or Metastatic Salivary Gland Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Renato Martins, Principal Investigator, University of Washington
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 7674; NCI-2012-00892 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2012-06-05; First posted 2012-06-07 (Estimated); Results first posted 2018-08-10 (Actual); Last update posted 2018-09-28 (Actual); Status verified 2018-08

CONDITIONS: Recurrent Salivary Gland Cancer; Stage IVA Salivary Gland Cancer; Stage IVB Salivary Gland Cancer; Stage IVC Salivary Gland Cancer
MeSH Terms: conditions — Salivary Gland Neoplasms | interventions — eribulin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment (eribulin mesylate) (Experimental): Patients receive eribulin mesylate IV over 2-5 minutes on days 1 and 8. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: eribulin mesylate

INTERVENTIONS:
Drug: eribulin mesylate — Given IV
  Other Names: B1939; E7389; ER-086526; halichrondrin B analog

SUMMARY:
Researchers are doing a research study to examine the use of eribulin (eribulin mesylate) in patients with salivary gland cancer. Researchers want to know if eribulin is safe and effective in treating salivary gland cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Evaluate the response rate of eribulin per Response Evaluation Criteria In Solid Tumors (RECIST) in patients with locally advanced refractory or metastatic salivary gland cancer (SGC).

SECONDARY OBJECTIVES:

I. Determine the safety and toxicity of eribulin in patients with locally advanced refractory or metastatic SGC.

II. Evaluate the duration of response and time-to-progression.

OUTLINE:

Patients receive eribulin mesylate intravenously (IV) over 2-5 minutes on days 1 and 8. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up at 30 days.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically or cytologically documented salivary gland cancers; patients that do not have a salivary gland primary must have one of the following histologies - adenoid cystic carcinoma, mucoepidermoid carcinoma, acinic cell carcinoma
* Patients must have recurrent and/or metastatic disease that is progressive and not amenable to surgery or curative radiotherapy occurring within 6 months of study entry, as evidenced by: at least a 20% increase in radiographically or clinically measurable disease, appearance of any new lesions, or deterioration in clinical status
* Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1, or 2
* Patients with measurable disease per RECIST 1.1 criteria

  * At least one lesion of >= 1.5 cm in long-axis diameter for non lymph nodes or >= 1.5 cm in short-axis diameter for lymph nodes which is serially measurable according to RECIST 1.1 using either computerized tomography (CT) or magnetic resonance imaging (MRI)
  * Lesions that have had radiotherapy must show evidence of progressive disease (PD) based on RECIST 1.1 to be deemed a target lesion
* Absolute neutrophil count >= 1,500/μL
* Platelets >= 100,000/μL
* Creatinine clearance >= 40 mL/min
* Bilirubin =< 1.5 upper limit of normal (ULN)
* Alkaline phosphatase =< 3 ULN; if total ALP is > 3 x ULN (in the absence of liver metastasis) or > 5 x ULN in subjects with liver metastasis AND the subject is known to have bone metastases, then liver ALP iso-enzyme should be used to assess liver function rather than total ALP
* Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) =< 3 X ULN
* Women of child-bearing potential (WOCP) and men must agree to use adequate contraception (hormonal or barrier method of birth control or abstinence) prior to study entry and for the duration of study participation
* Life expectancy of > 12 weeks
* Signed and dated informed consent document indicating that the patient has been informed of all the pertinent aspects of the trial prior to enrollment

Exclusion Criteria:

* Patients with symptomatic central nervous system (CNS) metastases must have stable disease after treatment with surgery or radiation therapy
* Second primary malignancy that is clinically detectable or clinically significant at the time of consideration for study enrollment
* Radiotherapy within 14 days of study treatment
* Major surgery within 21 days of study treatment; minor surgery within 2 weeks of study treatment; placement of vascular access device and biopsies allowed and is not considered major or minor surgery
* Treatment with any chemotherapy or investigational agents within 4 weeks of the start of study treatment; subjects must have recovered from toxicities of prior therapy
* Patients with peripheral neuropathy >= grade 2
* Significant cardiovascular impairment: congestive heart failure > class II according to the New York Heart Association (NYHA), unstable angina or myocardial infarction within 6 months of enrollment, or serious cardiac arrhythmia (> grade 2)
* Concomitant severe or uncontrolled medical disease
* Significant psychiatric or neurologic disorder which would compromise participation in the study
* Pregnant or breast-feeding females

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2012-05-08 (Actual); Primary Completion 2017-08-23 (Actual); Study Completion 2017-08-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Renato Martins, MD, MPH, Principal Investigator — Fred Hutchinson Cancer Research Center/University of Washington Cancer Consortium
Locations (1):
- Fred Hutchinson Cancer Research Center/University of Washington Cancer Consortium, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Seattle Cancer Care Alliance/University of Washington Phase II open label study enrolled patients at a single site between May 2012 and August 2015.
Pre-assignment Details: Twenty-nine patients were consented and treated.
Groups:
- Treatment (Eribulin Mesylate): Eribulin mesylate (1.4 mg/m2) administered intravenously (IV) over 2-5 minutes on days 1 and 8 of a 21 day cycle. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.
Period: Overall Study
Arm/Group | Treatment (Eribulin Mesylate)
Started | 29
Completed | 29
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Baseline participant measures are based on total eligible, consented and treated patients.
Groups:
- Treatment (Eribulin Mesylate): Patients receive Eribulin mesylate (1.4 mg/m2) administered intravenously (IV) over 2-5 minutes on days 1 and 8 of a 21 day cycle. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.
Arm/Group | Treatment (Eribulin Mesylate)
Number analyzed (Participants) | 29
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 15
  >=65 years | 14
Age, Continuous [Median (Full Range); unit: years] | 63 [23 to 79]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 20
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 28
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 26
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 29

OUTCOME MEASURES:

1. Primary Outcome: Response Rate
Description: Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1) for target lesions and assessed by either CT or MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR, summarized using frequencies and percentages.
Time Frame: From date of first study therapy until date of first documented disease progression or date of death from any cause, unacceptable toxicity or withdrawal of patient consent, whichever occurred first, assessed up to 36 days post last dose of study therapy.
Population: All participants receiving at least 1 dose of study intervention and at least 1 assessment post-baseline.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Eribulin Mesylate)
Number analyzed (Participants) | 29
Participants
  Complete Response (CR) | 1
  Partial Response (PR) | 2
  Stable Disease (SD) | 23
  Progressive Disease (PD) | 3

2. Secondary Outcome: Duration of Tumor Response (Complete (CR) and Partial (PR) Response Only)
Description: Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1) for target lesions and assessed by either CT or MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR, reported as median values.
Time Frame: as for outcome 1
Population: Participants receiving at least 1 dose of study intervention and at least 1 assessment post-baseline who achieved a CR or PR per RECIST 1.1.
Measure: Median (Full Range); unit: weeks
Arm/Group | Treatment (Eribulin Mesylate)
Number analyzed (Participants) | 3
weeks | 33.7 [24.0 to 77.9]

3. Secondary Outcome: Time to Progression
Description: Either 1. Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1) for target lesions and assessed by either CT or MRI: Progressive Disease (PD), > 20% increase in the sum of the longest diameter (SLD) target lesions taking as reference the smallest SLD recorded since the treatment started (nadir) and minimum 5 mm increase over the nadir; or 2. Radiographic progression per treating physician CT or MRI scan review.
Time Frame: From date of first study therapy until date of first documented disease progression or date of death from any cause, whichever occurred first, assessed up to 36 days post last dose of study therapy.
Population: All participants receiving at least 1 dose of study intervention and at least 1 assessment post-baseline. Does not include 7 patients taken off study before radiological progression: Toxicity = 3, Clinical PD = 4.
Measure: Median (Full Range); unit: Weeks
Arm/Group | Treatment (Eribulin Mesylate)
Number analyzed (Participants) | 22
Weeks | 18.0 [5.7 to 110.9]

4. Secondary Outcome: Disease Control Rate (DCR)
Description: Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1) for target lesions and assessed by either CT or MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Stable Disease (SD), neither sufficient shrinkage (compared to baseline) to qualify for partial or complete response (CR or PR) nor sufficient increase (taking as reference the smallest sum of diameters at baseline or while on study, whichever is smallest) to qualify for progressive disease (PD); Disease Control Rate (DCR) = CR + PR +SD.
Time Frame: as for outcome 1
Population: All participants receiving at least 1 dose of study intervention and at least 1 assessment post-baseline.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Eribulin Mesylate)
Number analyzed (Participants) | 29
Participants | 26

5. Secondary Outcome: Toxicity Rates
Description: Overall percentage of patients experiencing Grade 3 or higher toxicity, graded by National Cancer Institute (NCI) Common Toxicity Criteria Version 4.0
Time Frame: Adverse events collected from the time patient received the first dose of study therapy through 36 days following the last dose of study therapy or the start of a new cancer therapy, whichever occurred first, assessed up to 36 days post therapy.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Eribulin Mesylate)
Number analyzed (Participants) | 29
Participants | 14

ADVERSE EVENTS:
Time Frame: Adverse events collected from the time patient received the first dose of study therapy through 36 days following the last dose of study therapy or the start of a new cancer therapy, whichever occurred first, assessed up to 36 days post therapy.
Description: Any adverse events leading to a treatment interruption or dose reduction along with all adverse events that are grade 3 and higher were recorded.
Arm/Group | Treatment (Eribulin Mesylate)
All-Cause Mortality (participants affected / at risk) | 0/29
Serious Adverse Events (participants affected / at risk) | 3/29
Other Adverse Events (participants affected / at risk) | 16/29
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Eribulin Mesylate) (N=29)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1)
Pathological spinal fracture (Musculoskeletal and connective tissue disorders) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Eribulin Mesylate) (N=29)
Fatigue (General disorders) | 4 (4)
Malaise (General disorders) | 2 (2)
Creatinine increased (Investigations) | 2 (2)
Neutrophil count decreased (Investigations) | 8 (14)
Peripheral sensory neuropathy (Nervous system disorders) | 7 (10)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-02-14): https://cdn.clinicaltrials.gov/large-docs/68/NCT01613768/Prot_SAP_000.pdf